CLINICAL TRIAL: NCT06172010
Title: Rifampicin Combination Therapy Versus Targeted Antimicrobial Monotherapy in the Oral Antimicrobial Treatment Phase of Staphylococcal Prosthetic Joint Infection
Brief Title: Rifampicin Combination Therapy Versus Monotherapy for Staphylococcal Prosthetic Joint Infection
Acronym: RiCOTTA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: University Medical Center Groningen (Other); Onze Lieve Vrouwe Gasthuis (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Frisius Medisch Centrum (Other); Isala (Other); Martini Hospital Groningen (Other); Radboud University Medical Center (Other); Sint Maartenskliniek (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Erasmus Medical Center (Other); Alrijne Hospital (Other); Spaarne Gasthuis (Other); Reinier Haga Orthopedisch Centrum (Other); Tergooi Hospital (Other); Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Mark de Boer MD PhD, Prof dr MGJ de Boer, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-501620-26-00
Record Dates: First submitted 2023-11-23; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Prosthetic-joint Infection; Infection Hip; Infection; Knee, Joint
Keywords: rifampicin; clindamycin; levofloxacin; prosthetic joint infection; antimicrobial treatment
MeSH Terms: conditions — Infections | interventions — Clindamycin; Rifampin; Levofloxacin

STUDY DESIGN:
Intervention Model Description: randomized controlled open label trial with a non-inferiority design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral rifampicin-based combination therapy (Active Comparator): rifampicin 450mg BID + levofloxacin 500mg BID in the oral treatment phase with a total duration of antibiotics of 12 weeks
  Interventions: Drug: Rifampicin and levofloxacin
- Oral monotherapy with clindamycin (Experimental): clindamycin 600mg TID in the oral treatment phase with a total duration of antibiotics of 12 weeks
  Interventions: Drug: Clindamycin

INTERVENTIONS:
Drug: Clindamycin — antimicrobial treatment in oral treatment phase of staphylococcal prosthetic joint infection
  Arms: Oral monotherapy with clindamycin
Drug: Rifampicin and levofloxacin — antimicrobial treatment in oral treatment phase of staphylococcal prosthetic joint infection
  Arms: Oral rifampicin-based combination therapy

SUMMARY:
In this Dutch multicenter clinical trial, patients with a staphylococcal prosthetic joint infection, will, in the oral antibiotic treatment phase, be randomized between clindamycin monotherapy and rifampicin / levofloxacin combination therapy. The clinical endpoint will be treatment success one year after finishing antimicrobial treatment.

DETAILED DESCRIPTION:
This is a pragmatic, multicenter, randomized controlled open label trial with a non-inferiority design, comparing the efficacy of rifampicin-based combination antimicrobial therapy versus antimicrobial monotherapy with clindamycin during the oral treatment phase of prosthetic joint infection caused by Staphylococcus spp. The total duration of follow-up will be 15 months from the initial DAIR.

All adult patients, aged 18 years or older, diagnosed and hospitalized with hip- or knee PJI caused by Staphylococcus spp and treated by the DAIR strategy (see Interventions), are eligible for inclusion. The diagnosis of PJI is defined according to the EBJIS 2021 criteria. Exclusion criteria are a contra-indication for rifampicin (due to a resistant strain, a proven allergic reaction, difficult drug-drug-interactions or other contra-indications as listed in the SmPC's of the antibiotics), a contra-indication for levofloxacin and clindamycin and cotrimoxazole and tetracyclines (due to a resistant strain, a proven allergic reaction, difficult drug-drug-interactions or other contra-indications as listed in the SmPC's of the antibiotics), (iii)complicated S. aureus bacteremia or concurrent endocarditis requiring long-term iv antibiotic treatment > 3 weeks , (iv) an infection for which there are no suitable antibiotic choices to permit randomization between the two arms of the trial (for instance, where organisms are only sensitive to intravenous antibiotics), (v) treatment failure before the start of oral therapy, (vi) more than two separate surgical debridements , (vii)an unsatisfactory response to initial treatment leading to continuation of intravenous therapy beyond day 21, (viii) patients with an expected life expectancy <12 months, (ix) patients with a tumor prosthesis , (x) patients receiving chemotherapy for active malignancy in the next 12 months, (xi) patients who are scheduled in advance for chronic suppressive antibiotic therapy after the initial 12 weeks of antibiotic treatment, (xii) The patient is unlikely to comply with trial requirements following randomization in the opinion of the investigator, (xiii) Pregnancy or breastfeeding, (xiv) Patients who are not able to read or communicate in Dutch or English will be excluded from participating in this study.

The main trial endpoint is treatment success 15 months after DAIR (=1 year after finishing antibiotic treatment). Treatment success will be defined as absence of all of the following:

(I) Infection related re-surgery of the initially affected prosthetic joint (II) New antibiotic treatment for suspected or proven infection of the index joint.

(III) Ongoing use of antibiotics for the index joint at the end of follow-up. (IV) Death

Secondary outcomes are (a) Quality of life, measured with the 5-level EQ-5D version (EQ-5D-5L) questionnaires. The EQ-5D-5L is a standardized and validated measure of health status developed by the EuroQol Group to provide a comprehensive generic measure of health for clinical and economic appraisal. This 'quality of life' questionnaire will be scored at the time of randomization, at week 6 after the initial surgical debridement and after 3 months.

(b) Adverse events. The number of SAEs during antimicrobial treatment and follow up ii. The number of switches to a different oral regimen, iii. The number of antibiotic associated AEs (classified by the modified Hartwig and Siegel scale). (c) The number of patients developing Clostridioides difficile infection during treatment. (d) The occurrence of rifampicin resistance in bacteria in patients with a microbiologically confirmed failure of treatment.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Confirmed staphylococcal prosthetic hip or knee joint infection according to the current EBJIS 2021 definition of PJI
* The causative agents are (or include) S. aureus or and/or Coagulase-negative staphylococci (CNS)
* Treatment is according to the DAIR-procedure

Exclusion Criteria:

(i) a contra-indication for rifampicin (e.g. a resistant strain or proven allergic reaction or difficult drug-drug-interactions) (ii) complicated S. aureus bacteremia or concurrent endocarditis requiring long-term iv antibiotic treatment > 2 weeks (iii) An infection for which there are no suitable antibiotic choices to permit Randomization between the two arms of the trial (for instance, where organisms are only sensitive to intravenous antibiotics) (iv) treatment failure before the start of oral therapy, (v) an unsatisfactory response to initial treatment leading to continuation of intravenous therapy beyond day 21, (vi) patients with an expected life expectancy <12 months, (vii) patients with a tumor prosthesis (viii) patients receiving chemotherapy for active malignancy in the next 12 months (ix) patients who are scheduled in advance for chronic suppressive antibiotic therapy for >12 months, (x) The patient is unlikely to comply with trial requirements following Randomization in the opinion of the investigator (xi) Pregnancy (xii) Patients who are not able to read or communicate in Dutch or English will be excluded from participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
treatment success | 15 months after DAIR
  Proportion of patients with treatment success 15 months after DAIR (=1 year after finishing antibiotic) in both randomised groups treatment). Treatment success will be defined as absence of all of the following: (I) Infection related re-surgery of the initially affected prosthetic joint (II) New antibiotic treatment for suspected or proven infection of the index joint.
  (III) Ongoing use of antibiotics for the index joint at the end of follow-up. (IV) Death

SECONDARY OUTCOMES:
Quality of life of patients at baseline and after 6 and 12 weeks | at the time of randomization, at week 6 after surgical debridement and after 3 months.
  Quality of life, measured with the 5-level EQ-5D version (EQ-5D-5L) questionnaires. The number and percentage of patients reporting each level of problem on each dimension of the EQ-5D-5L will be decribed.
Adverse events | through study completion, an average of 15 months
  The number of (S)AEs during antimicrobial treatment and follow up (including mortality).
  ii. The proportion of patients switching to a different oral regimen in both study arms iii. The proportion of patient with antibiotic side effects (classified by the modified Hartwig and Siegel scale) in both study arms iv. The proportion of patient developing Clostridioides difficile infection during treatment in both study arms v. The proportion of patient with rifampicin resistance in bacteria in patients with a microbiologically confirmed failure of treatment in both study arms.
Development of new rifampicin resistance | through study completion, an average of 15 months
  The proportion of patients developing rifampicin resistance in patients with a confirmed microbiological relapse with the same micro-organism in both study arms

CONTACTS AND LOCATIONS:
Overall Officials: Henk Scheper, MD, Study Director — LUMC
Locations (13):
- Netherlands (13):
  - LUMC, Leiden, Zuid Hollans
  - Amsterdam UMC, Amsterdam
  - OLVG, Amsterdam
  - Martini ziekenhuis, Groningen
  - UMCG, Groningen
  - Spaarne gasthuis, Hoofddorp
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Alrijne Ziekenhuis, Leiderdorp
  - Radboud UMC, Nijmegen
  - Sint maartenskliniek, Nijmegen
  - Erasmus MC, Rotterdam
  - Elisabeth Tweesteden Ziekenhus, Tilburg
  - Stichting Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scheper H, Gerritsen LM, Pijls BG, Van Asten SA, Visser LG, De Boer MGJ. Outcome of Debridement, Antibiotics, and Implant Retention for Staphylococcal Hip and Knee Prosthetic Joint Infections, Focused on Rifampicin Use: A Systematic Review and Meta-Analysis. Open Forum Infect Dis. 2021 Jul 1;8(7):ofab298. doi: 10.1093/ofid/ofab298. eCollection 2021 Jul. PMID 34258321
- See also: Website with information for patients and physicians about RiCOTTA study — http://www.protheseinfectie.nl